CLINICAL TRIAL: NCT01519726
Title: CYP3A4 Metabolism Before and After Surgery Induced Weight Loss in Morbidly Obese Patients Using Midazolam as a Model Drug
Brief Title: CYP3A4 Metabolism Before and After Surgery Induced Weight Loss Using Midazolam as Model Drug
Acronym: MEMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Catherijne Knibbe, Professor in Pharmacology, Hospital pharmacist, St. Antonius Hospital
Other Study IDs: MEMO study
Record Dates: First submitted 2012-01-04; First posted 2012-01-27 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Midazolam

ARMS (1):
- Morbidly obese patients (Experimental)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam

SUMMARY:
Before and during bariatric surgery patients are given oral and i.v. midazolam, respectively and blood samples are drawn to establish midazolam time-concentration profiles. After 0.5-2 years, and substantial weight loss, oral and i.v. midazolam are administered once more and blood samples are taken again.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40
* undergoing bariatric surgery

Exclusion Criteria:

* use of drug inducing or inhibiting CYP3A4 activity
* pregnancy, breastfeeding
* renl insufficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Difference in midazolam clearance in morbidly obese patients before and 0.5-2 years after surgery | 0.5-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Hospital, Nieuwegein, Netherlands